CLINICAL TRIAL: NCT00960375
Title: Randomized Trial of a Smoking Cessation Program for Persons With SMI
Brief Title: Smoking Cessation for Veterans With Severe and Persistent Mental Illness
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURA-001-09S
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Schizoaffective Disorder; Schizophrenia; Affective Psychosis, Bipolar; Affective Disorders, Psychotic
Keywords: smoking cessation; serious mental illness
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder; Affective Disorders, Psychotic; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BTSCS (Experimental): BTSCS lasts 3 months, includes two 60-minute group meetings per week (24 group meetings total), and is delivered in small groups of 4-8 participants run by a trained interventionist. BTSCS includes: (1) An individual motivational enhancement meeting during the first week of treatment to help participants think about individual reasons for smoking cessation; (2) Breath carbon monoxide monitoring and goal-setting at the beginning of each meeting; (3) Skills for reducing smoking; (4) Social Skills Training; (5) Education about the biology of SPMI and smoking and the physiological harm caused by smoking; (5) Relapse prevention training; (6) Education about and assistance with nicotine replacement therapy for participants who are interested in learning about and trying it.
  Interventions: Behavioral: BTSCS
- StSST (Active Comparator): The StSST program is adapted from a 9-session weekly smoking cessation group program developed at the Outpatient Research Program of the Maryland Psychiatric Research Center and designed for people with schizophrenia. In this study, the StSST program meet twice per week for 3 months (24 sessions total). Participants complete a breath carbon monoxide test at the start of each group meeting. StSST groups provide education about smoking and support for quitting.
  Interventions: Behavioral: StSST

INTERVENTIONS:
Behavioral: BTSCS — BTSCS lasts 3 months, includes two 60-minute group meetings per week (24 group meetings total), and is delivered in small groups of 4-8 participants run by a trained interventionist. BTSCS includes: (1) An individual motivational enhancement meeting during the first week of treatment to help participants think about individual reasons for smoking cessation; (2) Breath carbon monoxide monitoring and goal-setting at the beginning of each meeting; (3) Skills for reducing smoking; (4) Social Skills Training; (5) Education about the biology of SPMI and smoking and the physiological harm caused by smoking; (5) Relapse prevention training; (6) Education about and assistance with nicotine replacement therapy for participants who are interested in learning about and trying it.
  Arms: BTSCS
Behavioral: StSST — The StSST program is adapted from a 9-session weekly smoking cessation group program developed at the Outpatient Research Program of the Maryland Psychiatric Research Center and designed for people with schizophrenia. In this study, the StSST program meet twice per week for 3 months (24 sessions total). Participants complete a breath carbon monoxide (CO) test at the start of each group. StSST groups provide education about smoking and support for quitting.
  Arms: StSST

SUMMARY:
The investigators have developed an intervention called Behavioral Treatment of Smoking Cessation in SPMI (BTSCS), an innovative intervention that supplements pharmacotherapy and education with contingency management and a multifaceted behavioral group treatment program that lasts for three months (24 group meetings). BTSCS is designed to address the cognitive, motivational, and social support problems characteristic of people with SPMI.

The investigators propose to conduct a randomized trial for persons with SPMI that compares (1) BTSCS: a 6-month manualized smoking cessation program adapted from an effective substance abuse treatment program for this population to (2) StSST: a standard manualized smoking cessation program which reflects current best practices.

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable death in the United States. Smoking contributes to increased rates of diseases such as lung cancer and heart disease, and adds dangerous complications to health problems such as diabetes and obesity. Despite widespread recognition of the devastating health effects of smoking, over 70% of people with schizophrenia and other serious and persistent mental illnesses (SPMI) smoke cigarettes, a rate that is at least double that of the general population and remains high despite decreases in rates of smoking in the general population. These extraordinary smoking rates contribute to elevated morbidity and mortality, have other life-threatening health-related consequences, and increase health care costs for treating smoking related illnesses in this population. Treating smoking is critical in improving the health of people with SPMI.

The newly revised VA/Department of Defense Clinical Practice Guideline for the Management of Tobacco Use outlines the VHA's comprehensive program for smoking cessation. Beginning in 1997, the VA central office directed that the Agency for Health Care Policy and Research (AHCPR) smoking cessation guideline (the 5 A's - Ask, Advise, Assess, Assist, Arrange) be implemented in all its health care facilities. Reinforcing their commitment to increasing veterans' access to evidence-based smoking cessation interventions, the VHA recently released a new policy mandating that smoking cessation treatment be made available without restriction at all VA sites. Our previous study implementing the 5A's in community mental health clinics has found reduced smoking and increased use of smoking cessation aids such as nicotine replacement therapy (NRT), but no only modest increases in abstinence. Implementation of the 5 A's was limited by inability to adequately assist patients to stop smoking. Consideration of how best to supplement the "Assist" and "Arrange" phases reveals the troubling observation that existing "best practice" treatments for smoking cessation have limited effectiveness for persons with SPMI. The most widely tested treatments consist generally of adaptations of American Lung Association (ALA) or comparable 10-14 session weekly groups supplemented by either nicotine replacement therapy (NRT) or Bupropion. Such programs produce low abstinence rates (0-25%) at end of intervention. Sustained abstinence is virtually non-existent. Abstinence at 6-month or 1-year follow-up points ranges from 0-10%.

We have developed an intervention the treatment of cocaine and heroin use disorders among persons with SPMI, called Behavioral Treatment for Substance Abuse in Serious and Persistent Mental Illness (BTSAS). BTSAS was developed with a series of National Institute on Drug Abuse (NIDA-funded treatment development grants as a treatment program for substance abuse that accommodated the cognitive and motivational impairments that characterize SPMI. The goal was to incorporate strategies that have been found to be effective in reducing drug use more generally, but to tailor them to meet the needs of people with SPMI. BTSAS provides a model for this application's test of an innovative smoking cessation treatment. Our basic premise is that we must first acknowledge nicotine dependence as an addiction with characteristics common to other substance addictions, and then specify the additional biological, social, cognitive, psychological and environmental barriers to quitting smoking for people with SPMI. We must then fully optimize available technologies for addiction in general and smoking cessation in particular to address these deficits. Existing approaches to smoking cessation for persons with SPMI do not use the full range of biological, contingency management, social modeling and behavioral tools that have been shown to work in treating other addictions in this population. Further, research on treatment of substance use disorders in persons with SPMI has suggested that, for best outcomes, interventions may need to be more intensive that what is provided for other groups of substance abusers. Applied to smoking, this suggests that for people with SPMI, smoking cessation may need to be more intensive than the 9 weekly sessions typical of conventional smoking cessation programs.

Based on our work developing BTSAS, and the above features of smoking in SPMI, we have developed an intervention called Behavioral Treatment of Smoking Cessation in SPMI (BTSCS), an innovative intervention that supplements pharmacotherapy and education with breath carbon monoxide monitoring and a multifaceted behavioral group treatment program that lasts for three months (24 sessions). BTSCS is designed to address the cognitive, motivational, and social support problems characteristic of people with SPMI. We propose to conduct a randomized clinical trial comparing BTSCS to a standard smoking cessation treatment.

Specific Aims: To determine if BTSCS is more effective in producing abstinence from smoking than a manualized smoking cessation program that reflects current best practices (StSST).

Hypothesis 1: BTSCS will result in greater rates of abstinence than StSST as shown by:

1. A higher percentage of negative expired carbon monoxide levels at biweekly treatment sessions
2. Increased days of abstinence reported at biweekly treatment sessions
3. A higher percentage of negative expired carbon monoxide levels immediately post-treatment.
4. A higher percentage of participants reporting abstinence in the 7-day interval preceding the post-treatment assessment.

Secondary Aims: We will assess the effectiveness of BTSCS on a set of intermediate outcomes including a reduction in smoking severity and improvement in readiness to quit smoking among smokers who have not been able to quit. We will also assess if increased treatment attendance and use of NRT's and bupropion moderate the hypothesized increases in abstinence.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of severe and persistent mental illness (SPMI) including a diagnosis of a psychotic disorder in keeping with criteria established by the Serious Mental Illness Treatment Research and Evaluation Center (SMITREC) -Schizophrenic disorders, affective psychoses and other psychotic diagnoses. We also include individuals with a diagnosis of Major Depression with psychotic features and PTSD.
* Age 18-75
* Nicotine dependence as defined by a score of 5 or higher on the Fagerstrom Tolerance Scale OR Participants who currently smoke at least 10 cigarettes per day
* Participants will not meet criteria for current alcohol/substance dependence (other than nicotine)
* Willingness ability to provide consent to participate.

Exclusion Criteria:

* Documented history of severe neurological disorder or severe head trauma with loss of consciousness
* Severe or profound mental retardation by chart review.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2010-04; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie E Bennett, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland

REFERENCES:
- [Derived] Bennett ME, Brown CH, Li L, Himelhoch S, Bellack A, Dixon L. Smoking Cessation in Individuals With Serious Mental Illness: A Randomized Controlled Trial of Two Psychosocial Interventions. J Dual Diagn. 2015;11(3-4):161-73. doi: 10.1080/15504263.2015.1104481. PMID 26457385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants attended outpatient mental health programs at the Baltimore, Perry Point, and Washington DC VA Medical Centers. Participants had DSM-IV diagnoses of schizophrenia spectrum disorders, affective psychosis, other psychotic disorder, major depression with psychotic features, or post-traumatic stress disorder.
Pre-assignment Details: To ensure functional impairment in line with SMI, participants with PTSD had to have worked less than 25% of the past year or receive disability payment for PTSD.
Groups:
- BTSCS: BTSCS includes two 60-minute groups/week (24 total). It is delivered in groups of 4-8 participants run by a trained interventionist. It includes: (1) individual motivational enhancement session to help participants think about personal reasons for change; (2) Breath CO monitoring and goal-setting; (3) Skills for reducing smoking; (4) Social Skills Training; (5) Education about negative health effects of smoking; (5) Relapse prevention; (6) Education about and assistance with nicotine replacement therapy.
- StSST: The StSST program was adapted from a 9-session weekly smoking cessation group program developed at the Outpatient Research Program of the Maryland Psychiatric Research Center and designed for people with schizophrenia. In this study, the StSST program meets twice per week for 3 months (24 sessions total). Participants will complete a breath CO test at the start of each education session with no associated feedback of results or financial contingency. To avoid possible discussion of the CO test and results, participants will do the CO test individually just outside the group room. There is no payment or contingency for CO testing in this condition. StSST groups will provide education about smoking and support for quitting. Smoking education sessions will involve weekly (24 sessions total) smoking cessation educational groups modeled after Addington et al. (1998) and modified using the educational materials of the American Cancer Society (ACS) Fresh Start Program.
Period: Overall Study
Arm/Group | BTSCS | StSST
Started | 92 | 87
Completed | 72 | 65
Not Completed | 20 | 22
Not completed — Lost to Follow-up | 20 | 22

BASELINE CHARACTERISTICS:
Population: 179 participants were randomized: 92 to BTSCS and 87 to StSST.
Groups:
- BTSCS: BTSCS lasts 3 months, includes two 60-minute group sessions per week (24 sessions total), and is delivered in small groups of 4-8 participants run by a trained therapist. BTSCS includes the following: (1) An individual motivational enhancement session during the first week of treatment to help participants think about individual reasons for smoking cessation; (2) Contingency management and goal-setting at the beginning of each session; (3) Skills for reducing smoking; (4) Social Skills Training; (5) Education about the biology of SPMI and smoking and the physiological harm caused by smoking; (5) Relapse prevention training; (6) Education about and assistance with nicotine replacement therapy for participants who are interested in learning about and trying it.
- Total: Total of all reporting groups
Arm/Group | BTSCS | StSST | Total
Number analyzed (Participants) | 92 | 87 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (13.0) | 54.1 (7.0) | 54.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 19
  Male | 77 | 83 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 90 | 87 | 177
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 65 | 62 | 127
  White | 23 | 17 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 92 | 87 | 179

OUTCOME MEASURES:

1. Primary Outcome: Number of Cigarettes Smoked Per Day
Description: Number of cigarettes smoked per day for the last 7 days
Time Frame: day
Population: All randomized
Measure: Mean (Standard Deviation); unit: number of cigarettes
Arm/Group | BTSCS | StSST
Number analyzed (Participants) | 92 | 87
number of cigarettes | 15.4 (9.8) | 14.9 (10.0)
Statistical Analysis 1: Comparison: BTSCS vs StSST; Smoking reduction outcomes were examined in the randomized sample using data from baseline and post-treatment assessments. The variable examined was self-reported number of cigarettes smoked per day during the last 7 days. This variable was skewed so a natural log transformation was applied before linear mixed model analysis; Test type: Superiority or Other; p = 0.489, ANOVA

2. Primary Outcome: Abstinence From Tobacco
Description: Self-reported abstinence from tobacco + breath CO < 10 ppm
Time Frame: 7 days
Population: All randomized to condition
Measure: Number; unit: participants
Arm/Group | BTSCS | StSST
Number analyzed (Participants) | 92 | 87
participants | 10 | 6
Statistical Analysis 1: Comparison: BTSCS vs StSST; This outcome was examined in the randomized sample. Abstinence was defined as self-reported no smoking in the last 7 days + expired CO ≤ 10 PPM. To assess difference in change between conditions, we tested the significance of the condition-by-time interaction using repeated measured mixed models with a random participant effect. Time was binary: post-treatment versus baseline. We used a logistic model for binary outcomes; Test type: Superiority or Other; p = 0.685, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant for the duration of their study participation (9 months).
Description: Adverse events were reported to the IRB yearly.
Groups:
- StSST: The StSST program is adapted from a 9-session weekly smoking cessation group program developed at the Outpatient Research Program of the Maryland Psychiatric Research Center and designed for people with schizophrenia. In this study, the StSST program meets twice per week for 3 months (24 sessions total). Participants will complete a breath CO test at the start of each education session with no associated feedback of results or financial contingency. To avoid possible discussion of the CO test and results, participants do the CO test individually just outside the group room. There is no payment or contingency for CO testing in this condition. StSST groups provide education about smoking and support for quitting. Smoking education groups involve weekly (24 groups total) smoking cessation educational groups modeled after Addington et al. (1998) and modified using the educational materials of the American Cancer Society (ACS) Fresh Start Program.
Arm/Group | BTSCS | StSST
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/87
Other Adverse Events (participants affected / at risk) | 0/92 | 0/87

LIMITATIONS AND CAVEATS:
The sample was mostly male, African-American, and recruited at VAMCs; it is unclear if findings would generalize to community settings. Many declined to participate; the sample represents persons with SMI who are interested in quitting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No